CLINICAL TRIAL: NCT02444806
Title: The Clinical Effectiveness of PSG Versus Limited Respiratory Polygraphy During NIV Set up in COPD-OSA Overlap Syndrome: A Randomised Controlled Trial
Brief Title: PSG Versus Oxim-capnography to Setup Home NIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14/LO/2088
Record Dates: First submitted 2015-05-12; First posted 2015-05-15 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: COPD; OSA
Keywords: Sleep disordered breathing; Domiciliary NIV
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Full Polysomnography (Active Comparator): Patients will have NIV settings established using overnight full polysomnography.
  Interventions: Other: Full polysomnography
- Oximetry-capnography (Active Comparator): Patients will have NIV settings established using only Oximetry-capnography and subjective sleep comfort.
  Interventions: Other: Oximetry-capnography

INTERVENTIONS:
Other: Full polysomnography — Full sleep and respiratory monitoring with EEG
  Other Names: Polysomnography
  Arms: Full Polysomnography
Other: Oximetry-capnography — Limited monitoring with nurse observation and continuous oximetry-capnography overnight for NIV titration.
  Other Names: Limited respiratory monitoring
  Arms: Oximetry-capnography

SUMMARY:
The study aims to compare 2 different strategies used to setup non-invasive ventilation in patients with OCPD-OSA overlap.

DETAILED DESCRIPTION:
With limited comparative data to support the different strategies, there is substantial variation across Europe and the United States in the methods used by clinicians to set up home non-invasive ventilation (NIV) for patients with chronic respiratory failure as a consequence of sleep disordered breathing. Indeed with few data to support the practice, many centres employ full montage polysomnography, which is not only a significant physical burden to the patient but also a financial burden to the healthcare provider in terms of the facilities required, staff training and equipment.

The investigators propose to undertake a randomised controlled trial to compare the clinical effectiveness, in terms of the change in daytime arterial partial pressure of carbon dioxide (PaCO2) at 3 months, of limited respiratory polygraphy and full polysomnography to set up NIV in patients with COPD-OSA overlap. Secondary outcome measures at 3 months will include overnight control of gas exchange, subjective sleep quality, health related quality of life and ventilator adherence. COPD-OSA overlap are a patient group that have a rising prevalence with limited data currently available detailing NIV set up, which wholly supports the rationale of using this increasingly important group as a target population for this trial.

ELIGIBILITY:
Inclusion Criteria:

* COPD (as defined by GOLD criteria[4])
* OSA (ODI > 7.5 events/hr, AHI > 5events/hr)
* PaCO2 > 6 kPa
* BMI > 30 kg/m2

Exclusion Criteria:

* Decompensated respiratory failure (pH < 7.35)
* Inability to tolerate NIV (< 4 hours usage at in hospital titration)
* Contraindication to NIV
* Pregnancy
* Aged <18
* Significant physical or psychiatric co-morbidity that would prevent compliance with trial protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
PaCO2 (Arterial blood gas analysis) | 3 months
  Arterial blood gas analysis

SECONDARY OUTCOMES:
Health related quality of life (CAT, SRI) | 3 months
  CAT, SRI
Spirometry (FEV1, FVC) | 3 months
  FEV1, FVC
Subjective sleep comfort (VAS) | 3 months
  VAS
Objective sleep comfort (Actigraphy) | 3 months
  Actigraphy
Respiratory mechanics (to include, work of breathing, PEEPdyn, Cdyn, EMGdi, EMGpara) | Day 1
  Invasive respiratory mechanics performed on discharge NIV settings to include, work of breathing, PEEPdyn, Cdyn, EMGdi, EMGpara
NIV compliance (machine recorded) | 3 months
  NIV machine recorded compliance

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Patout M, Arbane G, Cuvelier A, Muir JF, Hart N, Murphy PB. Polysomnography versus limited respiratory monitoring and nurse-led titration to optimise non-invasive ventilation set-up: a pilot randomised clinical trial. Thorax. 2019 Jan;74(1):83-86. doi: 10.1136/thoraxjnl-2017-211067. Epub 2018 Mar 30. PMID 29602814